CLINICAL TRIAL: NCT04243161
Title: Respiratory Muscle Training in Patients With Spinal Cord Injury
Brief Title: RMT in Patients With Spinal Cord Injury
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of time
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PR(AG)26/2018
Record Dates: First submitted 2020-01-20; First posted 2020-01-28 (Actual); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Spinal Cord Injuries
Keywords: Spinal Cord Injury; Rehabilitation; Respiratory Muscle Training; Quality of Life
MeSH Terms: conditions — Spinal Cord Injuries | interventions — High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Common clinical practice (pulmonary expansion exercises, drainage of secretions and training of inspiratory muscles) + expiratory muscle training at 50% load after MIP measurement.
  Interventions: Other: Experimental
- Group 2 (Active Comparator): Common clinical practice (pulmonary expansion exercises, drainage of secretions and training of inspiratory muscles) + expiratory muscle training at 30% load after MIP measurement.
  Interventions: Other: Control

INTERVENTIONS:
Other: Experimental — The study variables PIM, PEM, FVC, PEF and EQ-5D quality of life questionnaire will be measured on the first day when patient incorporated into the seating position in the patient's bed. Reassessments will be performed every two week till patient discharge from hospital. After that patient will be assessed after 4 month and 1 year after the SCI.
  SCIM III will be administered at discharge, 4 month later and 1 year after the injury.
  Common clinical practice (pulmonary expansion exercises,drainage of secretions and training of inspiratory muscles) + expiratory muscle training at 50% load after MIP measurement.
  The intensity of the treatment will be 50% of the PIM and PEM value (increasing the load in 2 cmH2O weekly). Three sets of 10 reps will be performed, with one total of 30 repetitions, resting 1 minute between each series.
  The sessions will be held once per day, from monday to friday, during the entire hospital admission.
  Other Names: High intensity training
  Arms: Group 1
Other: Control — The study variables PIM, PEM, FVC, PEF and EQ-5D quality of life questionnaire will be measured on the first day when patient incorporated into the seating position in the patient's bed. Reassessments will be performed every two week till patient discharge from hospital. After that patient will be assessed after 4 month and 1 year after the SCI.
  SCIM III will be administered at discharge, 4 month later and 1 year after the injury.
  Common clinical practice (pulmonary expansion exercises,drainage of secretions and training of inspiratory muscles) + expiratory muscle training at 30% load after MIP measurement.
  The intensity of the treatment will be 30% of the PIM value (increasing the load in 2 cmH2O weekly). Three sets of 10 reps will be performed, with one total of 30 repetitions, resting 1 minute between each series.
  The sessions will be held once per day, from monday to friday, during the entire hospital admission.
  Other Names: Usual intensity training
  Arms: Group 2

SUMMARY:
Spinal Cord Injury (SCI) is an involvement of the spinal cord, a nerve cord protected by the spine and extends from the base of the brain to the lumbar region. The spinal cord lesion causes complete or incomplete paralysis of voluntary mobility and absence, partial or total, of any sensitivity below the affected area; In addition, it also involves the lack of control over the sphincters of urination and intestinal evacuation, disorders of sexuality and fertility, alterations of the Vegetative Nervous System and risk of suffering other complications not less important as: bedsores, spasticity, kidney processes, ...

The cervical and dorsal cord injury severely affects respiratory function due to paralysis and deterioration of the respiratory muscles. Several types of respiratory muscle training (RMT) have been described to improve respiratory function for people with SCI in the literature.

Despite the relatively small number of studies included in this review, the meta-analysis of the pooled data indicates that RMT would be effective in increasing respiratory muscle strength and also lung volumes for people with SCI.

More research is needed to obtain functional results after EMR, such as dyspnea, cough efficacy, respiratory complications, hospital admissions due to respiratory complications and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acute spinal cord injury from C5 to T11 (AIS A-B)
* No tracheotomy user or invasive mechanical ventilation.
* Age between 18 years - 75 years.

Exclusion Criteria:

* Not wanting to participate in the study.
* Not meet inclusion criteria
* Cognitive or psychiatric disorder that does not allow you to participate in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximum respiratory pressures (PIM and PEM) | Through study completion, an average of 1 year
  Measured with respiratory pressure gauge
  Assessments:
  Baseline, every two weeks while patient still admitted in hospital, after 4 month and after 1 year.
Peak Cough Flow (PCF). | Through study completion, an average of 1 year
  Measured with a peak cough flow meter
  Assessments:
  Baseline, every two weeks while patient still admitted in hospital, after 4 month and after 1 year.
Forced Spirometry (FVC). | Through study completion, an average of 1 year
  Measured with a spirometer
  It is the maximum volume of exhaled air, with the maximum possible effort, starting from a maximum inspiration. It is expressed as volume (in ml) and is considered normal when it is greater than 80% of its theoretical value.
  Assessments:
  Baseline, every two weeks while patient still admitted in hospital, after 4 month and after 1 year.
Peak expiratory Flow (PEF) | Through study completion, an average of 1 year
  Measured with a spirometer
  It is the Maximum Flow (Peak expiratory Flow Right--(PEF)) that can be generated during a forced expiration maneuver; Measurement in liters per second.
  Baseline, every two weeks while patient still admitted in hospital, after 4 month and after 1 year.

SECONDARY OUTCOMES:
Measurement of independence in spinal cord injury and respiratory function | Through study completion, an average of 1 year
  Measured with SCIM III Test
  Assessments:
  Baseline, hospital discharge, after 4 month and after 1 year.
Quality of life questionnaire (EQ-5D). | Through study completion, an average of 1 year
  Measured with EuroQuol 5-D test
  Its a subjective test which goes from 0 to 100 in quality of life perception.
  Assessments:
  Baseline, hospital discharge, after 4 month and after 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Bernat Planas Pascual, PT, MSc, Principal Investigator — Hospital Universitari Vall d'Hebron Research Institute
Locations (1):
- Hospital Universitari Vall d'Hebron Research Institute, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gohl O, Walker DJ, Walterspacher S, Langer D, Spengler CM, Wanke T, Petrovic M, Zwick RH, Stieglitz S, Glockl R, Dellweg D, Kabitz HJ. [Respiratory Muscle Training: State of the Art]. Pneumologie. 2016 Jan;70(1):37-48. doi: 10.1055/s-0041-109312. Epub 2016 Jan 20. German. PMID 26789431
- [Result] Mitchell MD, Yarossi MB, Pierce DN, Garbarini EL, Forrest GF. Reliability of surface EMG as an assessment tool for trunk activity and potential to determine neurorecovery in SCI. Spinal Cord. 2015 May;53(5):368-74. doi: 10.1038/sc.2014.171. Epub 2014 Dec 2. PMID 25448189
- [Result] Postma K, Haisma JA, Hopman MT, Bergen MP, Stam HJ, Bussmann JB. Resistive inspiratory muscle training in people with spinal cord injury during inpatient rehabilitation: a randomized controlled trial. Phys Ther. 2014 Dec;94(12):1709-19. doi: 10.2522/ptj.20140079. Epub 2014 Jul 31. PMID 25082923
- [Result] Tamplin J, Berlowitz DJ. A systematic review and meta-analysis of the effects of respiratory muscle training on pulmonary function in tetraplegia. Spinal Cord. 2014 Mar;52(3):175-80. doi: 10.1038/sc.2013.162. Epub 2014 Jan 14. PMID 24418958
- [Result] Galeiras Vazquez R, Rascado Sedes P, Mourelo Farina M, Montoto Marques A, Ferreiro Velasco ME. Respiratory management in the patient with spinal cord injury. Biomed Res Int. 2013;2013:168757. doi: 10.1155/2013/168757. Epub 2013 Sep 9. PMID 24089664
- [Result] Terson de Paleville D, McKay W, Aslan S, Folz R, Sayenko D, Ovechkin A. Locomotor step training with body weight support improves respiratory motor function in individuals with chronic spinal cord injury. Respir Physiol Neurobiol. 2013 Dec 1;189(3):491-7. doi: 10.1016/j.resp.2013.08.018. Epub 2013 Aug 31. PMID 23999001
- [Result] Berlowitz DJ, Tamplin J. Respiratory muscle training for cervical spinal cord injury. Cochrane Database Syst Rev. 2013 Jul 23;2013(7):CD008507. doi: 10.1002/14651858.CD008507.pub2. PMID 23881660